CLINICAL TRIAL: NCT01435746
Title: A Randomized, Controlled Pilot Trial of Transfusion Requirements After Orthotopic Liver
Brief Title: Transfusion Requirements After Orthotopic Liver Transplantation
Acronym: TROLL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients could be recruited for this study
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karsten Gavenis, Dr., University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TROLL11
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Anemia
Keywords: liver transplantation; intensive care; red blood cell transfusion
MeSH Terms: conditions — Anemia | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liberal Transfusion (Experimental): Patients in the liberal transfusion group will receive red blood cell transfusions when their hemoglobin concentration drops below 10 g/dl. The aim should be to reach a hemoglobin concentration between 10 and 12 g/dl.
  Interventions: Behavioral: Red blood cell transfusion
- Conservative Transfusion (Active Comparator): Patients in the conservative transfusion group will receive red blood cell transfusions when their hemoglobin concentration drops below 8 g/dl. The aim should be to reach a hemoglobin concentration between 8 and 10 g/dl.
  Interventions: Behavioral: Red blood cell transfusion

INTERVENTIONS:
Behavioral: Red blood cell transfusion — The intervention of this trial is the regime of red blood cell transfusion. The control group will receive red blood cell transfusions according to a conservative regime, whereas the experimental group will receive red blood cell transfusion according to a liberal transfusion regime.

SUMMARY:
The objective of this trial is to evaluate different transfusion strategies in patients after liver transplantation. Patients in the experimental arm will be given red blood cell (RBC) transfusion according to a liberal strategy, i. e., transfusions should be given, when hemoglobin concentration falls below 10 g/dl, and hemoglobin concentration should be maintained between 10 and 12 g/dl. Patients in the control arm will be given red blood cell (RBC) transfusion according to a restrictive strategy, i. e., transfusions should be given, when hemoglobin concentration falls below 8 g/dl, and hemoglobin concentration should be maintained between 8 and 10 g/dl.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver transplantation
* Patients considered to have euvolemia after initial treatment by attending physicians

Exclusion Criteria:

* Patients age 18 or less
* Patients undergoing combined liver-kidney transplantation
* Patients requiring renal replacement therapy before liver transplantation for longer than two weeks
* Inability to receive blood products
* Patient with active blood loss at the time of enrollment
* Pregnancy
* Imminent death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Composite of death, graft loss and renal failure | 30 days after randomization

SECONDARY OUTCOMES:
Renal function | 30 days after randomization
  Renal function will be assessed by estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany